CLINICAL TRIAL: NCT00168324
Title: A Study of the Safety and Efficacy of a New Treatment for Macular Edema Resulting From Retinal Vein Occlusion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 206207-008
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2009-08-26 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Dexamethasone; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 700 µg Dexamethasone (Experimental): 700 µg dexamethasone intravitreal implant administered on Day 0 and Day 180.
  Interventions: Drug: 700 µg Dexamethasone
- 350 µg Dexamethasone followed by 700 µg Dexamethasone (Experimental): 350 µg dexamethasone intravitreal implant administered on Day 0 and 700 µg dexamethasone intravitreal implant on Day 180.
  Interventions: Drug: 700 µg Dexamethasone; Drug: 350 µg Dexamethasone
- Sham Injection followed by 700 µg Dexamethasone (Sham Comparator): Sham injection on Day 0 and 700 µg dexamethasone intravitreal implant on Day 180.
  Interventions: Drug: 700 µg Dexamethasone; Other: Sham Injection

INTERVENTIONS:
Drug: 700 µg Dexamethasone — 700 µg dexamethasone intravitreal implant administered on Day 0 and/or Day 180.
  Other Names: Posurdex®
Drug: 350 µg Dexamethasone — 350 µg Dexamethasone intravitreal implant administered on Day 0.
  Other Names: Posurdex®
  Arms: 350 µg Dexamethasone followed by 700 µg Dexamethasone
Other: Sham Injection — Sham injection on Day 0.
  Arms: Sham Injection followed by 700 µg Dexamethasone

SUMMARY:
This study will evaluate the safety and efficacy of an intravitreal implant of dexamethasone for the treatment of macular edema associated with retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with macular edema resulting from retinal vein occlusion
* Decrease in visual acuity in at least one eye as a result of macular edema (20/50 or worse)
* Visual acuity in other eye no worse than 20/200

Exclusion Criteria:

* Known anticipated need for ocular surgery within next 12 months
* History of glaucoma or current high eye pressure requiring more than 1 medication
* Diabetic retinopathy
* Uncontrolled systemic disease
* Known steroid-responder
* Use of systemic steroids
* Use of warfarin/heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2004-10-01 (Actual); Primary Completion 2008-03-01 (Actual); Study Completion 2008-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (13):
- Los Angeles, California, United States
- Sydney, Australia
- Graz, Austria
- Halifax, Nova Scotia, Canada
- Brno, Czechia
- Créteil, France
- Karlsruhe, Germany
- Rehovot, Israel
- Tabacalera, Mexico
- Makati, Philippines
- Coimbra, Portugal
- Arcadia, South Africa
- Kaohsiung City, Taiwan

REFERENCES:
- [Background] Haller JA, Bandello F, Belfort R Jr, Blumenkranz MS, Gillies M, Heier J, Loewenstein A, Yoon YH, Jacques ML, Jiao J, Li XY, Whitcup SM; OZURDEX GENEVA Study Group. Randomized, sham-controlled trial of dexamethasone intravitreal implant in patients with macular edema due to retinal vein occlusion. Ophthalmology. 2010 Jun;117(6):1134-1146.e3. doi: 10.1016/j.ophtha.2010.03.032. Epub 2010 Apr 24. PMID 20417567

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomly assigned during the double-blind period of the study to treatment with 700 µg dexamethasone, 350 µg dexamethasone, or sham injection on Day 0. Patients who qualified to continue in the open-label period of the study received 700 µg dexamethasone on Day 180.
Period: Double-Blind Period
Arm/Group | 700 µg Dexamethasone | 350 µg Dexamethasone Followed by 700 µg Dexamethasone | Sham Injection Followed by 700 µg Dexamethasone
Started | 201 | 196 | 202
Completed | 189 | 189 | 189
Not Completed | 12 | 7 | 13
Period: Open-Label Period
Arm/Group | 700 µg Dexamethasone | 350 µg Dexamethasone Followed by 700 µg Dexamethasone | Sham Injection Followed by 700 µg Dexamethasone
Started | 164 (Not all patients who completed the double-blind period entered the open-label period.) | 155 (Not all patients who completed the double-blind period entered the open-label period.) | 158 (Not all patients who completed the double-blind period entered the open-label period.)
Completed | 160 | 147 | 152
Not Completed | 4 | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 700 µg Dexamethasone | 350 µg Dexamethasone Followed by 700 µg Dexamethasone | Sham Injection Followed by 700 µg Dexamethasone | Total
Number analyzed (Participants) | 201 | 196 | 202 | 599
Age, Customized [Number; unit: participants]
  <45 years | 9 | 7 | 9 | 25
  45-65 years | 83 | 84 | 90 | 257
  >65 years | 109 | 105 | 103 | 317
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 92 | 85 | 272
  Male | 106 | 104 | 117 | 327

OUTCOME MEASURES:

1. Secondary Outcome: Number of Patients With 15 or More Letter Improvement in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. The numbers of patients with at least a 15 or more letter improvement in BCVA in the study eye at each visit are presented.
Time Frame: Day 90, Day 180
Population: Intent-to-Treat: all randomized patients
Measure: Number; unit: Number of Participants
Groups:
- 700 µg Dexamethasone: 700 µg dexamethasone intravitreal implant administered on Day 0.
Arm/Group | 700 µg Dexamethasone | 350 µg Dexamethasone | Sham Injection
Number analyzed (Participants) | 201 | 196 | 202
Number of Participants
  Day 90 | 45 | 41 | 25
  Day 180 | 39 | 32 | 37

2. Secondary Outcome: Change From Baseline in Retinal Thickness in the Study Eye
Description: Retinal thickness is assessed by optical coherence tomography (OCT) in the study eye. The retina is the light-sensitive part of the eye. OCT is a laser-based, noninvasive, diagnostic system providing high-resolution, three-dimensional images of the retina. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Day 90, Day 180
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Microns (µm)
Arm/Group | 700 µg Dexamethasone | 350 µg Dexamethasone | Sham Injection
Number analyzed (Participants) | 201 | 196 | 202
Microns (µm)
  Baseline | 548.9 (185.45) | 541.6 (183.68) | 534.4 (187.38)
  Change from Baseline at Day 90 | -199.3 (194.54) | -144.1 (166.59) | -78.2 (150.05)
  Change from Baseline at Day 180 | -105.0 (197.83) | -91.4 (198.16) | -110.3 (175.59)

3. Primary Outcome: Cumulative Response Rate of 15 or More Letter Improvement
Description: The cumulative response rate of 15 or more letter improvement was based on the Kaplan-Meier estimate. A Kaplan-Meier analysis takes into account patients who dropped out from the study prior to achieving the 15 letter improvement. Values ranged from 0-1, with a higher number indicating a higher probability of response.
Time Frame: Up to 180 Days
Population: Intent-to-Treat: all randomized patients
Measure: Number; unit: Kaplan-Meier Estimate
Arm/Group | 700 µg Dexamethasone | 350 µg Dexamethasone | Sham Injection
Number analyzed (Participants) | 201 | 196 | 202
Kaplan-Meier Estimate
  Day 30 | 0.101 | 0.092 | 0.045
  Day 60 | 0.258 | 0.204 | 0.100
  Day 90 | 0.359 | 0.292 | 0.165
  Day 180 | 0.397 | 0.349 | 0.225

4. Secondary Outcome: Percentage of Patients With a Change From Baseline in BCVA by Category
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. Data are grouped into the following 5 categories based on change from baseline: ≥15 Letters Improvement, ≥5 and <15 Letters Improvement, No Change (Between -5 to +5 Letters), ≥5 and <15 Letters Worsening, and ≥15 Letters Worsening.
Time Frame: Baseline, Day 90
Population: Intent-to-Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | 700 µg Dexamethasone | 350 µg Dexamethasone | Sham Injection
Number analyzed (Participants) | 201 | 196 | 202
Percentage of Patients
  ≥15 Letters Improvement | 22.4 | 20.9 | 12.4
  ≥5 and <15 Letters Improvement | 39.8 | 42.3 | 34.2
  No Change (Between -5 to +5 Letters) | 27.4 | 23.5 | 34.7
  ≥5 and <15 Letters Worsening | 7.0 | 9.2 | 13.4
  ≥15 Letters Worsening | 3.5 | 4.1 | 5.4

5. Secondary Outcome: Percentage of Patients With a Change From Baseline in BCVA by Category
Description: as for outcome 4
Time Frame: Baseline, Day 180
Population: Intent-to-Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | 700 µg Dexamethasone | 350 µg Dexamethasone | Sham Injection
Number analyzed (Participants) | 201 | 196 | 202
Percentage of Patients
  ≥15 Letters Improvement | 19.4 | 16.3 | 18.3
  ≥5 and <15 Letters Improvement | 34.8 | 37.8 | 27.7
  No Change (Between -5 to +5 Letters) | 29.4 | 25.5 | 30.2
  ≥5 and <15 Letters Worsening | 10.9 | 10.7 | 14.9
  ≥15 Letters Worsening | 5.5 | 9.7 | 8.9

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) are reported for the double-blind treatment period through Month 6.
Description: The safety population included all randomized patients who received at least one dose of study medication and was used to assess AEs and SAEs.
Arm/Group | 700 µg Dexamethasone | 350 µg Dexamethasone | Sham Injection
Serious Adverse Events (participants affected / at risk) | 12/196 | 28/197 | 14/202
Other Adverse Events (participants affected / at risk) | 119/196 | 107/197 | 63/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 700 µg Dexamethasone (N=196) | 350 µg Dexamethasone (N=197) | Sham Injection (N=202)
Angina pectoris (Cardiac disorders) | 2 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 4 | 0
Intraocular pressure increased (Investigations) | 1 | 3 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 2 | 0
Syncope (Nervous system disorders) | 0 | 1 | 2
Glaucoma (Eye disorders) | 0 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Blindness (Eye disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Drowning (General disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 700 µg Dexamethasone (N=196) | 350 µg Dexamethasone (N=197) | Sham Injection (N=202)
Conjunctival haemorrhage (Eye disorders) | 39 | 35 | 26
Eye pain (Eye disorders) | 13 | 8 | 7
Maculopathy (Eye disorders) | 11 | 7 | 17
Conjunctival hyperaemia (Eye disorders) | 10 | 11 | 7
Intraocular pressure increased (Investigations) | 46 | 46 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.